CLINICAL TRIAL: NCT06695533
Title: "I Can Do This! Managing My Diabetes: A Pilot Project Using a Novel Word Game-based Workbook Intervention to Allow People Living With Diabetes to Increase Their Diabetes Self-efficacy"
Brief Title: I Can Do This! Managing My Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Center for Diabetes Translation Research (Other)
Responsible Party: Principal Investigator, Catherine Park, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008292; 2025P011698 (Other: Emory IRB)
Record Dates: First submitted 2024-11-16; First posted 2024-11-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
Keywords: Diabetes self-management; Patient education; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The workbook will be designed with the help of 5 focus group discussions. Five focus groups will include participants from one of the following categories: patients, caregivers, providers, and diabetes educators. Each focus group will have 6-10 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes self management (Experimental): Eligible participants will utilize the workbook for a span of 3 months
  Interventions: Behavioral: Diabetes self management workbook

INTERVENTIONS:
Behavioral: Diabetes self management workbook — The diabetes self-management workbook section used in this pilot study will focus on diet management, specifically carbohydrates, following ADA guidelines. It will include exercises based on the ADA diabetes plate method, aimed at helping subjects understand meal planning, food categories, portion sizes, goal setting, and the impact of foods on blood glucose levels. Activities will include word searches, crosswords, and goal-setting exercises. Subjects will begin the first section during a clinic visit. They can complete the workbook at home over three months, with input from subjects and Certified Diabetes Care and Education Specialists to refine the content.

SUMMARY:
The goals of this study are to:

1. Co-develop a user-friendly word game-based workbook format for patients with diabetes to understand how to manage their diabetes. For this study, the first section of the workbook will be developed to teach carbohydrate management.
2. Assess the feasibility and acceptability of the workbook.
3. Understand the implementation challenges that will be important for improving the workbook and preparing it for larger-scale effectiveness research.

Participants will be asked to:

* Complete the workbook during their waiting time in the clinic or at home.
* Engage in word games designed to teach diabetes management vocabulary and concepts.
* Attend follow-up sessions to assess changes in self-efficacy and glycemic control.

DETAILED DESCRIPTION:
Diabetes poses a significant public health challenge in the U.S., affecting approximately 37 million people, or 11% of the population. The prevalence is rising, particularly among youth, with a forecasted 700% increase in type 2 diabetes cases by 2060. Diabetes leads to severe health complications, including increased risks of heart attacks, strokes, and kidney failure, and affects nearly 1 million people worldwide with vision loss. Many individuals struggle to manage their diabetes effectively; only about 50% achieve proper glycemic control.

Diabetes self-management education is crucial for improving self-efficacy and adherence to treatment, yet only 5-7% of eligible patients receive this education. The American Diabetes Association advocates for individualized nutrition therapy, but access remains limited, especially for uninsured populations, exacerbating health disparities.

To address this gap, a novel word game-based workbook is proposed to enhance diabetes self-efficacy. This workbook can be used in waiting rooms or at home, offering an engaging way to learn about diabetes management through word games and puzzles. It aims to provide accessible education for underserved communities, improve glycemic control, and ultimately reduce diabetes-related disparities.

ELIGIBILITY:
Inclusion Criteria:

Focus group inclusion:

1. Patients: adult with diabetes and patient at the Midtown Clinic
2. Caregivers: partner, or caregiver of a patient with diabetes
3. Providers: Physician Assistant (PA), Nurse Practitioner (NP), or MD who cares for patients with diabetes
4. Diabetes educators: diabetes educator

Focus group exclusion:

1. Cannot speak/read English
2. Unwilling to participate in group discussion
3. Pregnancy

Aim 2 inclusion criteria:

1. Having type 2 diabetes which is not insulin dependent since insulin management adds another level of diabetes self-management that would confound self-efficacy scores.
2. Having a hemoglobin a1c less than 10% based on their last 3 hemoglobin a1c readings within the 2 years before the recruitment phase of the study. The ADA recommends the initiation of insulin therapy for individuals with a hemoglobin a1c above 10%, therefore the study will focus on an intervention for diabetes before insulin is likely to be part of the management plan.
3. Not having any conditions that could interfere with the accuracy of a hemoglobin a1c result: anemia, hemoglobinopathy, end-stage renal disease, chronic liver disease.
4. The ability to read a passage set at a fifth-grade literacy, a score of at least 3 on the Mini-Cog test scale which would represent a lower likelihood of dementia, and the ability to drive to medical visits.
5. Subjects will represent a diversity of age, educational level, and socioeconomic status (will use type of medical insurance as a proxy)

Aim 2 exclusion criteria:

1. Cannot speak/read English
2. Unwilling to return for a follow-up visit in 3 months
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes self-efficacy score (Diabetes management self-efficacy (DMSE) | Pre test, post test (3months)
  Measures the confidence of patients with diabetes regarding diet, exercise and medical treatment)
Knowledge of American Diabetes Association (ADA) diabetes plate method | Pre test, post test (3months)
  The ADA diabetes plate method is a meal planning tool that divides a plate into three sections: half for non-starchy vegetables, one-quarter for lean protein, and one-quarter for whole grains or starchy foods. It helps individuals with diabetes control portions and manage carbohydrate intake for better blood glucose control.
Acceptability of Intervention Measure (AIM) | Pre test, post test (3months)
  The Acceptability of Intervention Measure (AIM) is a tool used to assess how acceptable an intervention is to participants. The AIM is a 4-item instrument that uses a 5-point Likert scale
Feasibility of Intervention Measure (FIM) | Pre test, post test (3months)
  The Feasibility of Intervention Measure (FIM) is a tool used to assess the perceived feasibility of an intervention. The FIM is a 4-item instrument that uses a 5-point Likert scale.

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | Pre test, post test (3months)
  HbA1c, or glycated hemoglobin, measures average blood glucose levels over the past two to three months. It's expressed as a percentage, with higher values indicating poorer blood sugar control
Change in Weight | Pre test, post test (3months)
  Change in Weight over the course of study.
Change in Blood Pressure | Pre test, post test (3months)
  Change in Blood Pressure over the course of study.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Park, MD, Principal Investigator — Emory University; Saria Hassan, MD, Principal Investigator — Emory University
Locations (1):
- Emory Midtown Clinic, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-08-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT06695533/ICF_000.pdf